CLINICAL TRIAL: NCT01293162
Title: Study on the Role of a Combination of Nutraceuticals (Armolipid Prev) With an Effect on Blood Pressure and Lipids in the Control of Cardiovascular Risk
Brief Title: The Role of a Combination of Nutraceuticals in the Control of Cardiovascular Risk
Acronym: ARMOPREVCVR
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Bruno Trimarco, Full Professor of Cardiology, Federico II University
Other Study IDs: ARMOPREV-2011
Record Dates: First submitted 2011-02-09; First posted 2011-02-10 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic syndrome; Cardiovascular risk
MeSH Terms: conditions — Metabolic Syndrome | interventions — coenzyme Q10; Berberine; red yeast rice; policosanol; Folic Acid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- placebo
  Interventions: Drug: Armolipid Prev

INTERVENTIONS:
Drug: Armolipid Prev — Ortosiphon 300 mg/die, CoQ10 15 mg/die, Berberine 500 mg/die, red yeast 60 mg/die, policosanol 10 mg/die, Folic acid 200 mg/die
  Other Names: orthosiphon; CoQ10; berberine; red yeast; policosanol; folic acid

SUMMARY:
Cardiovascular risk has been shown to increase with increasing blood pressure values. As a consequence, it results mandatory to achieve lower blood pressure goals in all hypertensive patients, taking into account that all drugs always have some side effects that can be very dangerous and/or uncomfortable for the patients leading to a reduced compliance. Thus, pharmacological treatment should be delayed until it results really necessary.

The availability of natural substances with a therapeutic action has modified this scenario because of their reduced potential to cause undesirable effects (compared with drugs). In order to choose among various nutraceuticals (natural foods compounds with health benefits, including the prevention and/or treatment of diseases), preference should be given to those

* produced according to the same Good Manufacturing Practice used for drugs, to be sure that the finished product has a standard, reproducible composition
* for which efficacy and safety in the recommended indications are supported by clinical trials.

An example of a product with these characteristics is Armolipid Plus, a combination of nutraceuticals with a demonstrated anti-dyslipidaemic effect. Recently, a large clinical intervention study showed evidence that treatment with Armolipid Plus leads to a significant decrease in the overall cardiovascular risk, measured using the Framingham Risk Score.

Progress in Research and Development in this field has led to a new patented and registered combination of nutraceuticals: Armolipid Prev, containing orthosiphon and CoQ10, with antihypertensive activity, berberine, red yeast, policosanol and orthosiphon with antidyslipidaemic effect and folic acid, reducing plasma homocysteine levels.

In addition to the established anti-dyslipidaemic activity of Armolipid plus, Armolipid Prev has a significant antihypertensive effect, which is beneficial in all those patients with high blood pressure values without a defined indication to begin a pharmacological treatment according to the current guidelines. The antihypertensive effect of Armolipid Prev, documented by ambulatory blood pressure monitoring, in addition to the lowering effect on dyslipidaemia and even on abdominal girth, represents a new opportunity for complete and early, effective and safe cardiovascular disease prevention.

DETAILED DESCRIPTION:
Study on the role of a combination of nutraceuticals (Armolipid Prev) with an effect on blood pressure and lipids in the control of cardiovascular risk.

APv - cpr - 0210

1. Study rationale The strategies for the prevention of cardiovascular diseases always involve correction of wrong lifestyle habits, whereas use of pharmacological treatments is recommended only in patients with a high cardiovascular risk.

   This approach obviously leaves off a wide proportion of the population at low-moderate cardiovascular risk that could benefit from early BP-lowering treatment before development of organ damage or before it become irreversible, because in high-risk hypertensive patients, even intense cardiovascular therapy, through beneficial, is nonetheless unable to lower total cardiovascular risk below the high risk threshold.

   In the setting of cardiovascular prevention, presence of metabolic syndrome results particularly relevant, since it affects a large percentage of population and it has been demonstrated to increase the risk of cardiovascular events.

   However the mere lifestyle recommendations, despite useful, cannot always reach the established blood pressure and metabolic goals and reduce global cardiovascular risk.

   Moreover, cardiovascular risk has been shown to increase with increasing blood pressure values, so it results mandatory to achieve lower blood pressure goals, taking into account that all drugs always have some side effects that can be very dangerous and/or uncomfortable for the patients leading to a reduced compliance. Thus, pharmacological treatment should be started only if really necessary. The availability of natural substances with a therapeutic action has altered this scenario because of their reduced potential to cause undesirable effects (compared with drugs). In order to choose among various nutraceuticals (natural foods compounds with health benefits, including the prevention and/or treatment of diseases), preference should be given to those
   * produced according to the same Good Manufacturing Practice used for drugs, to be sure that the finished product has a standard, reproducible composition
   * for which efficacy and safety in the recommended indications are supported by clinical trials.

   An example of a product that meets these criteria is Armolipid Plus, a combination of nutraceuticals which allowed control of dyslipidaemia. Recently, a large clinical intervention study showed evidence that treatment with Armolipid Plus leads to a significant decrease in the overall cardiovascular risk, measured by the Framingham Risk Score.

   Progress in Research and Development in this field has led to a new patented and registered combination of nutraceuticals: Armolipid Prev, containing orthosiphon and CoQ10, with antihypertensive activity, berberine, red yeast, policosanol and orthosiphon with antidyslipidaemic effect and folic acid, reducing plasma homocysteine levels. In addition to the established anti-dyslipidaemic activity of Armolipid plus, Armolipid Prev has a significant antihypertensive effect, which is beneficial in all those patients with high blood pressure values without a defined indication to begin a pharmacological treatment according to the current guidelines. The antihypertensive effect of Armolipid Prev, documented by ambulatory blood pressure monitoring, in addition to the lowering effect on dyslipidaemia and even on abdominal girth, represents a new opportunity for complete and early, effective and safe cardiovascular disease prevention. In fact, in association with a balanced diet and healthy lifestyle, Armolipid Prev can encourage subjects to improve their lifestyle, thereby delaying the need for lipid-lowering drugs. Armolipid Prev is classified by the Ministry of Health as a food supplement in the Notification of 29th January 2010.
2. AIM OF THE STUDY

   Aim of the study is to evaluate the efficacy of a nutraceutical such as Armolipid Prev compared with simple advice on diet and a healthy lifestyle in:
   * achieving a greater reduction in the overall cardiovascular risk
   * reducing the incidence of metabolic syndrome
   * reducing the prevalence of microalbuminuria
   * reducing the prevalence of left ventricular hypertrophy evaluated on the ECG
   * increasing compliance to adopt a healthy lifestyle.
3. STUDY DESIGN Multicentre, randomized, controlled parallel-group study.
4. STUDY POPULATION At least 150 doctors will take part in the study; each will treat at least 10 subjects of both genders with diagnosis of metabolic syndrome and who require blood pressure control but without a defined indication to start a pharmacological treatment or in whom stable drug therapy did not achieve the established result.

   Indicators:

   GPs are required: 1) to record a full medical history, including smoking and drinking habits, based on a pre-defined clinical record; 2) to collect demographic and anthropometric measures (height, weight, waist circumference at the iliac crest); 3) to perform a complete physical exam.

   At the first visit and after 1, 3 and 12 months all eligible patients will perform a complete physical exam that includes measure of office blood pressure and heart rate in the sitting position and in triplicate, using a manual sphygmomanometer, according to international guidelines. Measurements will be rounded to the closest 2 mmHg interval.

   The baseline visit and the others screening visits also include examination of cell blood counts (CBCs), serum creatinine, sodium, potassium, uric acid, total cholesterol, triglycerides, HDL-cholesterol, glucose, GOT, GPT, CPK, urine analysis and microalbuminuria. LDL will be calculated starting from the total cholesterol, triglyceride and HDL-cholesterol.

   At the first visit and at the end of follow up all patients will be evaluated for the presence of Left Ventricular Hypertrophy by Electrocardiogram (ECG) and for cardiovascular risk assessment using Framingham cardiovascular risk score.

   Metabolic syndrome will be defined as the presence of at least 3 of the following 5 factors: increased blood pressure (≥ 130/85 and ≤ 140/90 mmHg); serum triglycerides ≥ 150 mg/dL; serum HDL cholesterol ≤ 40 mg/dL (males), ≤ 50 mg/dL (females); abdominal girth ≥ 104 cm (males), ≥ 88 cm (females); elevated fasting blood glucose ≥ 100 mg/dL.

   Hypertension will be defined according to 2003 ESH/ESC guidelines Diagnosis of Left Ventricular Hypertrophy will be assessed using the current ECG criteria (the Sokolow-Lyon index: S in V1 + R in V5 or V6 ≥ 35 mm and R in aVL ≥ 11 mm; the Cornell voltage criteria (S in V3 + R in aVL > 28 mm in men and S in V3 + R in aVL > 20 mm in women) at baseline and at the end of the follow-up.

   Cardiovascular risk will be calculated according to the Framingham risk score at baseline and at the end of the follow-up.

   The following will be excluded from the treatment: diabetics or hypertensive subjects with an indication for treatment, patients under lipid-lowering treatment and according to the Package Leaflet, all pregnant or breast-feeding women.

   Patients requiring cholesterol-lowering drug therapy, according to the international guidelines, will not be included in the study population.

   The primary endpoint is the improvement in the estimate of cardiovascular risk calculated by the FRS.

   Secondary endpoint:

   Reduction of incident metabolic syndrome Reduction in the prevalence of subjects with microalbuminuria Reduction in the prevalence of left ventricular hypertrophy on the ECG.

   4.1. Sample size

   According to results from a previous study performed on the efficacy of Armolipid Plus (-12% reduction in the FRS at 8 weeks compared with -6.5% with diet alone), an approximate estimate was made of the number of observations necessary so that the two percentages are significant at the 5% probability level: 600 cases in each group.
5. TREATMENTS all subjects will receive dietary counseling determined by the general practitioner depending on the subject's clinical condition, in accordance with the instructions of the Coordinating Site.

   Centralized randomization will be used to assign subjects to one of the two study treatments, placebo + diet or Armolipid Prev + diet.

   How Armolipid Prev will be taken 1 tablet daily of Armolipid Prev or placebo.

   Duration of treatment Subjects in both groups will take the assigned treatment for 12 months.
6. EVALUATION CRITERIA At the first visit and after 1, 3, 12 months blood pressure values and lipid profile will be assessed as well as the others clinical parameters necessary to evaluate the cardiovascular risk and to evaluate diagnosis of metabolic syndrome.

   In order to standardize the measurements, each doctor will be given a sphygmomanometer and a tape measure to estimate abdominal girth.
7. STUDY PROCEDURES Each doctor will initially be given a login and password allowing confidential and individual access to the website www.armolipid.net for data entry.

   The doctor will complete the appropriate form (also available on the armolipid.net site) and will assign the subject to one of two regimens: placebo + diet or Armolipid Prev + diet, based on what has been determined by centralised randomization under the responsibility of Prof. Bruno Trimarco.

   This procedure is undertaken by a telephone call to the Randomization Centre, which will automatically inform the doctor about the treatment to which the subject is to be assigned in order to keep a balanced ratio between the two groups. In order to avoid sampling errors, the doctor will include in the study the first 10 consecutive subjects who meet the admission criteria (see point 4).
8. STATISTICAL ANALYSIS The statistical analysis of baseline homogeneity will be undertaken using the chi-square test and analysis of variance, if appropriate.

   The statistical analysis to assess the clinical efficacy will be based on a comparison between differences at the various time points versus the baseline obtained in the two treatment groups and will be conducted using the chi-square test and analysis of variance, where appropriate.

   The level of significance will be considered to be an Alfa = 0.05 (type I error) and the power level a beta = 0.90 (type II error).
9. INSURANCE COVER This protocol is covered by an insurance policy taken out with AXA Assicurazioni e Investimenti, policy no.100720 (Milan Branch). The insurance will cover any injury to health sustained by patients and the economic damage arising from this, occurring during the period over which the policy is valid, which will be renewed on a year to year basis.
10. STUDY TIMELINES The study will start from the time the login and password have been delivered.
11. AVAILABILITY OF DATA All participants will be informed of the results once the data have been processed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of metabolic syndrome and requiring a blood pressure reduction without any indication to start a pharmacological therapy or in whom stable drug therapy has not achieved the desired results
* The presence of at least 3 of the following 5 factors:

  * increased blood pressure (≥ 130/85 and ≤ 140/90 mmHg)
  * serum triglycerides ³150 mg/dL
  * serum HDL cholesterol ≤ 40 mg/dL (males), ≤ 50 mg/dL (females)
  * abdominal girth ≥ 104 cm (males), ≥ 88 cm (females)
  * elevated fasting blood glucose ≥ 100 mg/dL

Exclusion Criteria:

* Diabetics or hypertensive subjects with an indication to start a pharmacological therapy
* Patients under lipid-lowering treatment
* Pregnant or breast-feeding women according to the Package Leaflet

Patients who require cholesterol-lowering drug therapy in accordance with the international guidelines will not be included in the study population

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Metabolic syndrome
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2010-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Cardiovascular risk | 12 months
  Reduction the global cardiovascular risk calculated according to Framingham risk score compared to baseline.
  Reduction of incident metabolic syndrome defined according to ATPIII criteria compared to baseline.
  Reduction of the prevalence of microalbuminuria evaluated by standard methods compared to baseline.
  Reduction of the prevalence of left ventricular hypertrophy evaluated by the ECG using the current ECG criteria (the Sokolow-Lyon index) compared to baseline.

SECONDARY OUTCOMES:
Life style | 12 months
  Increasing compliance with a healthy lifestyle assessed by office interview of the patients at baseline and at the end of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Trimarco, MD, Study Director — Federico II University, Dipartimento di medicina Clinica Scienze Cardiovascoalri ed Immunologiche
Locations (1):
- Ambulatorio Ipertensione e Unità Coronarica Federico II University, Napoli, Italy

REFERENCES:
- [Background] Izzo R, de Simone G, Giudice R, Chinali M, Trimarco V, De Luca N, Trimarco B. Effects of nutraceuticals on prevalence of metabolic syndrome and on calculated Framingham Risk Score in individuals with dyslipidemia. J Hypertens. 2010 Jul;28(7):1482-7. doi: 10.1097/HJH.0b013e3283395208. PMID 20498621
- See also: website of the High Blood Pressure Outpatient Clinic and UTIC of "Federico II" University of Naples — http://www.campaniasalute.com